CLINICAL TRIAL: NCT03827811
Title: Pharmacometrics to Advance Novel Regimens for Drug-resistant Tuberculosis
Brief Title: Pharmacometrics to Advance Novel Regimens for Drug-resistant Tuberculosis-PandrTB Tuberculosis
Acronym: PandrTB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cape Town (Other)
Collaborators: Partners in Health (Other); Epicentre (Other); Medecins Sans Frontieres, Netherlands (Other); Institute of Tropical Medicine, Belgium (Other); Interactive Research and Development (Other)
Responsible Party: Principal Investigator, Helen Margaret McIlleron, Professor, University of Cape Town
Other Study IDs: PandrTB
Record Dates: First submitted 2018-08-07; First posted 2019-02-01 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Multi-drug Resistant Tuberculosis
Keywords: MDR
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood will be stored for evaluation of genetic variants associated with drug concentrations and effects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PandrTB cohort: endTB and endTB-Q study participants on experimental regimen

SUMMARY:
PandrTB is a study of the pharmacokinetics(PK) and pharmacodynamics(PD) of bedaquiline, delamanid, clofazimine, linezolid, moxifloxacin, levofloxacin and pyrazinamide used in novel combinations to treat multidrug-resistant tuberculosis(MDR-TB).

DETAILED DESCRIPTION:
PandrTB is an observational study nested in the endTB (a randomized study that will evaluate five 9-month, injectable-sparing regimens) and endTB-Q (and RCT evaluating a 4 drug oral regimen given for 6 or 9 months) trials. These trials are providing evidence to support the transformation of MDR-TB treatment. As part of PandrTB: the plasma concentrations of the experimental arm drugs (the new and repurposed drugs bedaquiline, delamanid, clofazimine and linezolid, as well as levofloxacin, moxifloxacin and pyrazinamide) will be measured; MICs will be determined in baseline isolates; and MGIT cultures, additional to those in the endTB study, will be performed at weeks 6 and 10. Nonlinear mixed-effects models will describe the population PK of the drugs and a pharmacodynamic (PD) model of treatment response of Mycobacterium tuberculosis(Mtb) load over time. Recursive partitioning methods will evaluate baseline MICs and PK measures as drivers of treatment response (as described by the parameters of the PD model of initial treatment response of Mtb load over time, and the endTB trial endpoints: time to culture conversion, longer-term outcomes, and acquisition of phenotypic resistance). Thus the key drugs and plasma drug exposure thresholds for activity will be defined, and exposure-dependent synergy or antagonism identified. The risks of toxicities (as assessed in the endTB study) will be estimated, by plasma drug exposure and important comorbidity (including HIV infection). In this way, the PK-efficacy and PK-toxicity analyses will allow definition of target plasma drug exposures. Simulations will predict optimal doses. To advance the understanding of drug penetration, we will develop approaches to measure free drug plasma concentrations. Drug-drug interactions will be described. Thus PandrTB will inform how best to use these new and repurposed drugs in combination, to create the most effective and least toxic regimens while minimizing the development of further drug resistance.

ELIGIBILITY:
Inclusion Criteria:

All patients enrolled to the experimental arms of the endTB study and provide their written informed consent to participate in the PandrTB study.

Exclusion Criteria:

-

Ages: 15 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and adolescents (≥15 years) will be enrolled. There is increasing recognition that adolescents have been neglected in the development of treatments for diseases like HIV and TB, given that they comprise and important population. Minors are included in the endTB clinical trial and it would be wrong to exclude them from a PK study designed to optimize doses.
Sampling Method: Probability Sample
Enrollment: 625 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Drug exposure (AUC) | 5 years
  drug exposures derived using population PK models
Rate of decline of viable M.tubercolosis in sputum | 5 years
  A pharmacodynamic biomarker model of response to treatment will be used to derive the rate of decline of Mtb in MIGT cultures. The effect of PK on this measure will be evaluated.
Collecting adverse events as a measure of safety | 5 years
  The effect of pharmacokinetics on drug and regimen saftey will be evaluated using recursive partitioning methods.

CONTACTS AND LOCATIONS:
Overall Officials: Helen McIlleron, PhD, Principal Investigator — University of Cape Town
Locations (7):
- National Scientific Center of Phthisiopulmonology, Almaty, Kazakhstan
- Partners in Health Lesotho House 233 Corner Lancers and Caldwell Roads, Maseru, Lesotho
- Indus Hospital, Karachi, Pakistan
- Peru (2):
  - Peru-1, Lima
  - Peru_2, Lima
- Khayelitsha Town 2 Clinic, Cape Town, Western Cape, South Africa
- Hanoi Lung Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Horsburgh CR, Rusen ID, Mitnick CD. Optimizing MDR-TB clinical trials: insights from the first global MDR-TB Clinical Trials Landscape Meeting. Int J Tuberc Lung Dis. 2016 Dec 1;20(12):1-3. doi: 10.5588/ijtld.16.0568. No abstract available. PMID 28240564
- [Background] Diacon AH, Pym A, Grobusch MP, de los Rios JM, Gotuzzo E, Vasilyeva I, Leimane V, Andries K, Bakare N, De Marez T, Haxaire-Theeuwes M, Lounis N, Meyvisch P, De Paepe E, van Heeswijk RP, Dannemann B; TMC207-C208 Study Group. Multidrug-resistant tuberculosis and culture conversion with bedaquiline. N Engl J Med. 2014 Aug 21;371(8):723-32. doi: 10.1056/NEJMoa1313865. PMID 25140958
- [Background] Ahuja SD, Ashkin D, Avendano M, Banerjee R, Bauer M, Bayona JN, Becerra MC, Benedetti A, Burgos M, Centis R, Chan ED, Chiang CY, Cox H, D'Ambrosio L, DeRiemer K, Dung NH, Enarson D, Falzon D, Flanagan K, Flood J, Garcia-Garcia ML, Gandhi N, Granich RM, Hollm-Delgado MG, Holtz TH, Iseman MD, Jarlsberg LG, Keshavjee S, Kim HR, Koh WJ, Lancaster J, Lange C, de Lange WC, Leimane V, Leung CC, Li J, Menzies D, Migliori GB, Mishustin SP, Mitnick CD, Narita M, O'Riordan P, Pai M, Palmero D, Park SK, Pasvol G, Pena J, Perez-Guzman C, Quelapio MI, Ponce-de-Leon A, Riekstina V, Robert J, Royce S, Schaaf HS, Seung KJ, Shah L, Shim TS, Shin SS, Shiraishi Y, Sifuentes-Osornio J, Sotgiu G, Strand MJ, Tabarsi P, Tupasi TE, van Altena R, Van der Walt M, Van der Werf TS, Vargas MH, Viiklepp P, Westenhouse J, Yew WW, Yim JJ; Collaborative Group for Meta-Analysis of Individual Patient Data in MDR-TB. Multidrug resistant pulmonary tuberculosis treatment regimens and patient outcomes: an individual patient data meta-analysis of 9,153 patients. PLoS Med. 2012;9(8):e1001300. doi: 10.1371/journal.pmed.1001300. Epub 2012 Aug 28. PMID 22952439
- [Background] Dheda K, Esmail A, Limberis J, Maartens G. Selected questions and controversies about bedaquiline: a view from the field. Int J Tuberc Lung Dis. 2016 Dec 1;20(12):24-32. doi: 10.5588/ijtld.16.0065. PMID 28240569
- [Background] van Heeswijk RP, Dannemann B, Hoetelmans RM. Bedaquiline: a review of human pharmacokinetics and drug-drug interactions. J Antimicrob Chemother. 2014 Sep;69(9):2310-8. doi: 10.1093/jac/dku171. Epub 2014 May 23. PMID 24860154
- [Background] Gupta R, Wells CD, Hittel N, Hafkin J, Geiter LJ. Delamanid in the treatment of multidrug-resistant tuberculosis. Int J Tuberc Lung Dis. 2016 Dec 1;20(12):33-37. doi: 10.5588/ijtld.16.0125. PMID 28240570
- [Background] Lewis JM, Sloan DJ. The role of delamanid in the treatment of drug-resistant tuberculosis. Ther Clin Risk Manag. 2015 May 13;11:779-91. doi: 10.2147/TCRM.S71076. eCollection 2015. PMID 25999726
- [Background] Gler MT, Skripconoka V, Sanchez-Garavito E, Xiao H, Cabrera-Rivero JL, Vargas-Vasquez DE, Gao M, Awad M, Park SK, Shim TS, Suh GY, Danilovits M, Ogata H, Kurve A, Chang J, Suzuki K, Tupasi T, Koh WJ, Seaworth B, Geiter LJ, Wells CD. Delamanid for multidrug-resistant pulmonary tuberculosis. N Engl J Med. 2012 Jun 7;366(23):2151-60. doi: 10.1056/NEJMoa1112433. PMID 22670901
- [Background] O'Donnell MR, Padayatchi N, Metcalfe JZ. Elucidating the role of clofazimine for the treatment of tuberculosis. Int J Tuberc Lung Dis. 2016 Dec 1;20(12):52-57. doi: 10.5588/ijtld.16.0073. PMID 28240574
- [Background] Lamprecht DA, Finin PM, Rahman MA, Cumming BM, Russell SL, Jonnala SR, Adamson JH, Steyn AJ. Turning the respiratory flexibility of Mycobacterium tuberculosis against itself. Nat Commun. 2016 Aug 10;7:12393. doi: 10.1038/ncomms12393. PMID 27506290
- [Background] Van Deun A, Maug AK, Salim MA, Das PK, Sarker MR, Daru P, Rieder HL. Short, highly effective, and inexpensive standardized treatment of multidrug-resistant tuberculosis. Am J Respir Crit Care Med. 2010 Sep 1;182(5):684-92. doi: 10.1164/rccm.201001-0077OC. Epub 2010 May 4. PMID 20442432
- [Background] Tang S, Yao L, Hao X, Liu Y, Zeng L, Liu G, Li M, Li F, Wu M, Zhu Y, Sun H, Gu J, Wang X, Zhang Z. Clofazimine for the treatment of multidrug-resistant tuberculosis: prospective, multicenter, randomized controlled study in China. Clin Infect Dis. 2015 May 1;60(9):1361-7. doi: 10.1093/cid/civ027. Epub 2015 Jan 20. PMID 25605283
- [Background] U.S. Food and Drug Administration. NDA 204-384 Sirturo™ (bedaquiline 100 mg tablets) for the treatment of adults (≥ 18 years) as part of combination therapy of pulmonary multi-drug resistant tuberculosis (MDRTB). 2012 Nov 28;1-69
- [Background] Cox H, Ford N. Linezolid for the treatment of complicated drug-resistant tuberculosis: a systematic review and meta-analysis. Int J Tuberc Lung Dis. 2012 Apr;16(4):447-54. doi: 10.5588/ijtld.11.0451. PMID 22325685
- [Background] Nuermberger E. Evolving strategies for dose optimization of linezolid for treatment of tuberculosis. Int J Tuberc Lung Dis. 2016 Dec 1;20(12):48-51. doi: 10.5588/ijtld.16.0113. PMID 28240573
- [Background] Zvada SP, Denti P, Sirgel FA, Chigutsa E, Hatherill M, Charalambous S, Mungofa S, Wiesner L, Simonsson US, Jindani A, Harrison T, McIlleron HM. Moxifloxacin population pharmacokinetics and model-based comparison of efficacy between moxifloxacin and ofloxacin in African patients. Antimicrob Agents Chemother. 2014;58(1):503-10. doi: 10.1128/AAC.01478-13. Epub 2013 Nov 4. PMID 24189253
- [Background] Cox HS, Sibilia K, Feuerriegel S, Kalon S, Polonsky J, Khamraev AK, Rusch-Gerdes S, Mills C, Niemann S. Emergence of extensive drug resistance during treatment for multidrug-resistant tuberculosis. N Engl J Med. 2008 Nov 27;359(22):2398-400. doi: 10.1056/NEJMc0805644. No abstract available. PMID 19038891
- [Background] Cegielski JP, Dalton T, Yagui M, Wattanaamornkiet W, Volchenkov GV, Via LE, Van Der Walt M, Tupasi T, Smith SE, Odendaal R, Leimane V, Kvasnovsky C, Kuznetsova T, Kurbatova E, Kummik T, Kuksa L, Kliiman K, Kiryanova EV, Kim H, Kim CK, Kazennyy BY, Jou R, Huang WL, Ershova J, Erokhin VV, Diem L, Contreras C, Cho SN, Chernousova LN, Chen MP, Caoili JC, Bayona J, Akksilp S; Global Preserving Effective TB Treatment Study (PETTS) Investigators. Extensive drug resistance acquired during treatment of multidrug-resistant tuberculosis. Clin Infect Dis. 2014 Oct 15;59(8):1049-63. doi: 10.1093/cid/ciu572. Epub 2014 Jul 23. PMID 25057101
- [Background] Kang YA, Shim TS, Koh WJ, Lee SH, Lee CH, Choi JC, Lee JH, Jang SH, Yoo KH, Jung KH, Kim KU, Choi SB, Ryu YJ, Kim KC, Um S, Kwon YS, Kim YH, Choi WI, Jeon K, Hwang YI, Kim SJ, Lee HK, Heo E, Yim JJ. Choice between Levofloxacin and Moxifloxacin and Multidrug-Resistant Tuberculosis Treatment Outcomes. Ann Am Thorac Soc. 2016 Mar;13(3):364-70. doi: 10.1513/AnnalsATS.201510-690BC. PMID 26871879
- [Background] Johnson JL, Hadad DJ, Boom WH, Daley CL, Peloquin CA, Eisenach KD, Jankus DD, Debanne SM, Charlebois ED, Maciel E, Palaci M, Dietze R. Early and extended early bactericidal activity of levofloxacin, gatifloxacin and moxifloxacin in pulmonary tuberculosis. Int J Tuberc Lung Dis. 2006 Jun;10(6):605-12. PMID 16776446
- [Background] Gumbo T, Chigutsa E, Pasipanodya J, Visser M, van Helden PD, Sirgel FA, McIlleron H. The pyrazinamide susceptibility breakpoint above which combination therapy fails. J Antimicrob Chemother. 2014 Sep;69(9):2420-5. doi: 10.1093/jac/dku136. Epub 2014 May 12. PMID 24821594
- [Background] Andries K, Villellas C, Coeck N, Thys K, Gevers T, Vranckx L, Lounis N, de Jong BC, Koul A. Acquired resistance of Mycobacterium tuberculosis to bedaquiline. PLoS One. 2014 Jul 10;9(7):e102135. doi: 10.1371/journal.pone.0102135. eCollection 2014. PMID 25010492
- [Background] Pasipanodya JG, McIlleron H, Burger A, Wash PA, Smith P, Gumbo T. Serum drug concentrations predictive of pulmonary tuberculosis outcomes. J Infect Dis. 2013 Nov 1;208(9):1464-73. doi: 10.1093/infdis/jit352. Epub 2013 Jul 29. PMID 23901086
- [Background] Chigutsa E, Pasipanodya JG, Visser ME, van Helden PD, Smith PJ, Sirgel FA, Gumbo T, McIlleron H. Impact of nonlinear interactions of pharmacokinetics and MICs on sputum bacillary kill rates as a marker of sterilizing effect in tuberculosis. Antimicrob Agents Chemother. 2015 Jan;59(1):38-45. doi: 10.1128/AAC.03931-14. Epub 2014 Oct 13. PMID 25313213
- [Background] Modongo C, Pasipanodya JG, Magazi BT, Srivastava S, Zetola NM, Williams SM, Sirugo G, Gumbo T. Artificial Intelligence and Amikacin Exposures Predictive of Outcomes in Multidrug-Resistant Tuberculosis Patients. Antimicrob Agents Chemother. 2016 Sep 23;60(10):5928-32. doi: 10.1128/AAC.00962-16. Print 2016 Oct. PMID 27458224
- [Background] Srivastava S, Pasipanodya JG, Meek C, Leff R, Gumbo T. Multidrug-resistant tuberculosis not due to noncompliance but to between-patient pharmacokinetic variability. J Infect Dis. 2011 Dec 15;204(12):1951-9. doi: 10.1093/infdis/jir658. Epub 2011 Oct 21. PMID 22021624
- [Background] Drusano GL, Sgambati N, Eichas A, Brown DL, Kulawy R, Louie A. The combination of rifampin plus moxifloxacin is synergistic for suppression of resistance but antagonistic for cell kill of Mycobacterium tuberculosis as determined in a hollow-fiber infection model. mBio. 2010 Aug 10;1(3):e00139-10. doi: 10.1128/mBio.00139-10. PMID 20802826
- [Background] Chirehwa MT, Rustomjee R, Mthiyane T, Onyebujoh P, Smith P, McIlleron H, Denti P. Model-Based Evaluation of Higher Doses of Rifampin Using a Semimechanistic Model Incorporating Autoinduction and Saturation of Hepatic Extraction. Antimicrob Agents Chemother. 2015 Nov 9;60(1):487-94. doi: 10.1128/AAC.01830-15. Print 2016 Jan. PMID 26552972
- [Background] McIlleron H, Rustomjee R, Vahedi M, Mthiyane T, Denti P, Connolly C, Rida W, Pym A, Smith PJ, Onyebujoh PC. Reduced antituberculosis drug concentrations in HIV-infected patients who are men or have low weight: implications for international dosing guidelines. Antimicrob Agents Chemother. 2012 Jun;56(6):3232-8. doi: 10.1128/AAC.05526-11. Epub 2012 Mar 12. PMID 22411614
- [Background] Chigutsa E, Visser ME, Swart EC, Denti P, Pushpakom S, Egan D, Holford NH, Smith PJ, Maartens G, Owen A, McIlleron H. The SLCO1B1 rs4149032 polymorphism is highly prevalent in South Africans and is associated with reduced rifampin concentrations: dosing implications. Antimicrob Agents Chemother. 2011 Sep;55(9):4122-7. doi: 10.1128/AAC.01833-10. Epub 2011 Jun 27. PMID 21709081
- [Background] Savic RM, Ruslami R, Hibma JE, Hesseling A, Ramachandran G, Ganiem AR, Swaminathan S, McIlleron H, Gupta A, Thakur K, van Crevel R, Aarnoutse R, Dooley KE. Pediatric tuberculous meningitis: Model-based approach to determining optimal doses of the anti-tuberculosis drugs rifampin and levofloxacin for children. Clin Pharmacol Ther. 2015 Dec;98(6):622-9. doi: 10.1002/cpt.202. Epub 2015 Oct 22. PMID 26260983
- [Background] Shenje J, Ifeoma Adimora-Nweke F, Ross IL, Ntsekhe M, Wiesner L, Deffur A, McIlleron HM, Pasipanodya J, Gumbo T, Mayosi BM. Poor Penetration of Antibiotics Into Pericardium in Pericardial Tuberculosis. EBioMedicine. 2015 Sep 16;2(11):1640-9. doi: 10.1016/j.ebiom.2015.09.025. eCollection 2015 Nov. PMID 26870790
- [Background] Lenaerts A, Barry CE 3rd, Dartois V. Heterogeneity in tuberculosis pathology, microenvironments and therapeutic responses. Immunol Rev. 2015 Mar;264(1):288-307. doi: 10.1111/imr.12252. PMID 25703567
- [Background] Irwin SM, Prideaux B, Lyon ER, Zimmerman MD, Brooks EJ, Schrupp CA, Chen C, Reichlen MJ, Asay BC, Voskuil MI, Nuermberger EL, Andries K, Lyons MA, Dartois V, Lenaerts AJ. Bedaquiline and Pyrazinamide Treatment Responses Are Affected by Pulmonary Lesion Heterogeneity in Mycobacterium tuberculosis Infected C3HeB/FeJ Mice. ACS Infect Dis. 2016 Apr 8;2(4):251-267. doi: 10.1021/acsinfecdis.5b00127. Epub 2016 Feb 24. PMID 27227164
- [Background] Irwin SM, Gruppo V, Brooks E, Gilliland J, Scherman M, Reichlen MJ, Leistikow R, Kramnik I, Nuermberger EL, Voskuil MI, Lenaerts AJ. Limited activity of clofazimine as a single drug in a mouse model of tuberculosis exhibiting caseous necrotic granulomas. Antimicrob Agents Chemother. 2014 Jul;58(7):4026-34. doi: 10.1128/AAC.02565-14. Epub 2014 May 5. PMID 24798275
- [Background] Horita Y, Doi N. Comparative study of the effects of antituberculosis drugs and antiretroviral drugs on cytochrome P450 3A4 and P-glycoprotein. Antimicrob Agents Chemother. 2014 Jun;58(6):3168-76. doi: 10.1128/AAC.02278-13. Epub 2014 Mar 24. PMID 24663015
- [Background] Te Brake LH, Russel FG, van den Heuvel JJ, de Knegt GJ, de Steenwinkel JE, Burger DM, Aarnoutse RE, Koenderink JB. Inhibitory potential of tuberculosis drugs on ATP-binding cassette drug transporters. Tuberculosis (Edinb). 2016 Jan;96:150-7. doi: 10.1016/j.tube.2015.08.004. Epub 2015 Oct 9. PMID 26682943
- [Background] Svensson EM, Dooley KE, Karlsson MO. Impact of lopinavir-ritonavir or nevirapine on bedaquiline exposures and potential implications for patients with tuberculosis-HIV coinfection. Antimicrob Agents Chemother. 2014 Nov;58(11):6406-12. doi: 10.1128/AAC.03246-14. Epub 2014 Aug 11. PMID 25114140
- [Background] Svensson EM, Aweeka F, Park JG, Marzan F, Dooley KE, Karlsson MO. Model-based estimates of the effects of efavirenz on bedaquiline pharmacokinetics and suggested dose adjustments for patients coinfected with HIV and tuberculosis. Antimicrob Agents Chemother. 2013 Jun;57(6):2780-7. doi: 10.1128/AAC.00191-13. Epub 2013 Apr 9. PMID 23571542
- [Background] Pandie M, Wiesner L, McIlleron H, Hughes J, Siwendu S, Conradie F, Variava E, Maartens G. Drug-drug interactions between bedaquiline and the antiretrovirals lopinavir/ritonavir and nevirapine in HIV-infected patients with drug-resistant TB. J Antimicrob Chemother. 2016 Apr;71(4):1037-40. doi: 10.1093/jac/dkv447. Epub 2016 Jan 7. PMID 26747099
- [Background] Mallikaarjun S, Wells C, Petersen C, Paccaly A, Shoaf SE, Patil S, Geiter L. Delamanid Coadministered with Antiretroviral Drugs or Antituberculosis Drugs Shows No Clinically Relevant Drug-Drug Interactions in Healthy Subjects. Antimicrob Agents Chemother. 2016 Sep 23;60(10):5976-85. doi: 10.1128/AAC.00509-16. Print 2016 Oct. PMID 27458223
- [Background] Chigutsa E, Patel K, Denti P, Visser M, Maartens G, Kirkpatrick CM, McIlleron H, Karlsson MO. A time-to-event pharmacodynamic model describing treatment response in patients with pulmonary tuberculosis using days to positivity in automated liquid mycobacterial culture. Antimicrob Agents Chemother. 2013 Feb;57(2):789-95. doi: 10.1128/AAC.01876-12. Epub 2012 Nov 26. PMID 23183433
- [Background] Svensson E. A model-based analysis to describe bedaquiline's exposure-response relationship and predict the impact of drug-drug interactions. 9th Int workshop on Clinical Pharmacology of Tuberculosis Drugs 2016, Liverpool October 2016; Abstract O_01.
- [Background] Taubel J, Naseem A, Harada T, Wang D, Arezina R, Lorch U, Camm AJ. Levofloxacin can be used effectively as a positive control in thorough QT/QTc studies in healthy volunteers. Br J Clin Pharmacol. 2010 Apr;69(4):391-400. doi: 10.1111/j.1365-2125.2009.03595.x. PMID 20406223
- [Background] Naidoo A, Chirehwa M, McIlleron H, Naidoo K, Essack S, Yende-Zuma N, Kimba-Phongi E, Adamson J, Govender K, Padayatchi N, Denti P. Effect of rifampicin and efavirenz on moxifloxacin concentrations when co-administered in patients with drug-susceptible TB. J Antimicrob Chemother. 2017 May 1;72(5):1441-1449. doi: 10.1093/jac/dkx004. PMID 28175315
- See also: World Health Organization. Global tuberculosis report 2016. Geneva: WHO; 2016 — http://www.who.int/tb/publications/global_report/en/